CLINICAL TRIAL: NCT06755593
Title: Effectiveness of Intravenous Laser Therapy in Patients With Sciatica and Sleep Disorders at Binh Dinh Hospital of Traditional Medicine and Rehabilitation
Brief Title: Effectiveness of Intravascular Laser Therapy on Sleep Quality in Patients With Chronic Low Back Pain: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Le Hoang Minh Quan (Other)
Collaborators: Binh Dinh Hospital of Traditional Medicine and Rehabilitation (Unknown)
Responsible Party: Sponsor-Investigator, Le Hoang Minh Quan, Principal Investigator, University of Medicine and Pharmacy at Ho Chi Minh City
Organization: University of Medicine and Pharmacy at Ho Chi Minh City (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 445/QĐ-SYT
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Sleep Disorders; Sciatica
Keywords: sciatica; sleep disorders; intravenous laser; electroacupuncture
MeSH Terms: conditions — Sleep Wake Disorders; Sciatica | interventions — Electroacupuncture

STUDY DESIGN:
Intervention Model Description: A Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electroacupuncture and intravenous laser (Experimental): Participants in this group receive combined electroacupuncture and intravascular laser irradiation of blood (ILIB).
  * Electroacupuncture: Performed once daily for 10 consecutive days at a frequency of 60 Hz, 20 minutes per session. Acupuncture points include Jiaji (L3-S1), Dachangshu (BL25), Huantiao (GB30), Yinmen (BL37), Yanglingquan (GB34), Chengfu (BL36), Chengshan (BL57), and Kunlun (BL60).
  * Intravascular Laser Therapy: A sterile intravenous needle is inserted into a peripheral vein, and a laser fiber (630-650 nm, low-level laser) is introduced through the same entry site. The laser is connected to the laser source, delivering photobiomodulation for 30 minutes per session, 5 sessions per week, for 2 consecutive weeks (total 10 sessions).
  Intervention Name:
  * Procedure: Electroacupuncture
  * Device: Intravascular Low-Level Laser Therapy (ILIB)
  Interventions: Procedure: Electroacupuncture; Device: Intravascular Low-Level Laser Therapy (ILIB)
- Electroacupuncture (Active Comparator): Participants in this group receive electroacupuncture only.
  * Electroacupuncture: Performed once daily for 10 consecutive days, 20 minutes per session, using a frequency of 60 Hz.
  * Acupuncture Points: Jiaji (L3-S1), Dachangshu (BL25), Huantiao (GB30), Yinmen (BL37), Yanglingquan (GB34), Chengfu (BL36), Chengshan (BL57), and Kunlun (BL60).
  Intervention Name:
  - Procedure: Electroacupuncture
  Interventions: Procedure: Electroacupuncture

INTERVENTIONS:
Procedure: Electroacupuncture — Electroacupuncture is performed using sterile disposable acupuncture needles (0.30 × 25 mm) connected to an electroacupuncture stimulator (KWD808-1, Gujin Greatwall, China). Stimulation is applied at a frequency of 60 Hz for 20 minutes per session. Treatment is performed once daily for 10 consecutive days. Acupuncture points include Jiaji (L3-S1), Dachangshu (BL25), Huantiao (GB30), Yinmen (BL37), Yanglingquan (GB34), Chengfu (BL36), Chengshan (BL57), and Kunlun (BL60).
Device: Intravascular Low-Level Laser Therapy (ILIB) — Intravascular laser irradiation of blood (ILIB) is administered using a helium-neon laser device (Mini-630, 635 nm wavelength) manufactured by the Vietnam Laser Technology Center. A sterile optical fiber is inserted into a peripheral vein via a standard intravenous needle. The laser is connected to the fiber to deliver continuous photobiomodulation for 30 minutes per session, 5 sessions per week, for 2 consecutive weeks (10 sessions total). This device is used only in the experimental group in combination with electroacupuncture.
  Arms: Electroacupuncture and intravenous laser

SUMMARY:
Sciatica is a common condition worldwide, including in Vietnam, with prevalence rates ranging from 1.2% to 43%. Chronic sciatica is often associated with sleep disturbances, which can worsen pain perception and reduce quality of life. According to the 2023 report from the Binh Dinh Hospital of Traditional Medicine and Rehabilitation, sciatica accounted for approximately 26% of hospital admissions for musculoskeletal disorders.

Sleep disorders, particularly insomnia, are frequently reported among patients with chronic pain, forming a bidirectional relationship in which pain disrupts sleep, and poor sleep amplifies pain sensitivity. Current pharmacological treatments for insomnia often provide limited benefits and can lead to adverse effects with long-term use. Therefore, non-pharmacologic, integrative interventions have gained increasing interest.

Intravascular laser irradiation of blood (ILIB), also known as intravascular photobiomodulation, is a minimally invasive therapy that delivers low-level laser light (630-650 nm) directly into the venous circulation. ILIB has been reported to improve microcirculation, reduce oxidative stress, and modulate inflammation. Preliminary studies have suggested potential benefits for pain relief, sleep improvement, and functional recovery.

This randomized controlled pilot study aims to evaluate the effectiveness of intravascular laser therapy in improving sleep quality and pain among patients with chronic sciatica. Sixty-six participants will be randomly assigned to two groups:

* A control group receiving electroacupuncture, and
* An intervention group receiving intravascular laser therapy combined with electroacupuncture.

Treatment will be administered for 10 consecutive days. Clinical outcomes will be assessed using the Pittsburgh Sleep Quality Index (PSQI), Visual Analog Scale (VAS) for pain, Oswestry Disability Index (ODI), and Epworth Sleepiness Scale (ESS) at baseline, Day 7, and Day 15.

The study seeks to provide preliminary evidence supporting intravascular photobiomodulation as a safe, non-pharmacologic adjunct therapy for improving both pain and sleep quality in patients with chronic low back pain and sciatica.

DETAILED DESCRIPTION:
Sciatica, characterized by radiating pain along the sciatic nerve, is one of the most common causes of chronic low back pain. The condition affects approximately 13%-40% of adults globally and remains a major contributor to disability, reduced productivity, and impaired quality of life. In Vietnam, hospital-based surveys have reported that sciatica accounts for 12%-26% of inpatient admissions in traditional medicine and rehabilitation facilities.

Chronic musculoskeletal pain such as sciatica is frequently associated with sleep disorders. Studies indicate that up to 70% of patients with chronic pain experience poor sleep quality, and the relationship between pain and sleep is bidirectional: persistent pain interferes with sleep continuity, while sleep deprivation increases pain sensitivity and emotional distress. Conventional pharmacologic treatments for insomnia (such as benzodiazepines or non-benzodiazepine hypnotics) often provide temporary relief but may cause tolerance, dependence, or adverse cognitive effects. Consequently, non-pharmacologic and integrative approaches are increasingly emphasized in chronic pain management.

Intravascular photobiomodulation (ILIB), also referred to as intravascular laser irradiation of blood, is a minimally invasive technique that introduces low-level laser light (typically 630-650 nm) into the venous circulation. The photobiological effects of ILIB include enhanced oxygen transport, improved microcirculation, modulation of oxidative stress, and anti-inflammatory action. Clinical studies have demonstrated ILIB's potential in various chronic diseases, including musculoskeletal pain, vascular disorders, and metabolic dysfunctions. Preliminary evidence also suggests that ILIB may enhance sleep quality through regulation of circadian and autonomic function.

This randomized controlled pilot study was designed to evaluate the short-term efficacy of ILIB combined with electroacupuncture in improving pain and sleep quality in patients with chronic sciatica. The trial was conducted at the Binh Dinh Hospital of Traditional Medicine and Rehabilitation, Vietnam, from April to December 2024.

A total of 66 patients aged 18 years or older, diagnosed with chronic sciatica (pain duration ≥ 3 months) and sleep disturbance (Pittsburgh Sleep Quality Index > 5), were recruited and randomly assigned to one of two groups:

* Control Group (n = 33): Received electroacupuncture at 60 Hz for 20 minutes daily for 10 consecutive days, targeting Ashi points, Jiaji points (lumbar region), Dachangshu, Shangliao, and Ciliao.
* Intervention Group (n = 33): Received the same electroacupuncture regimen plus low-level intravascular laser irradiation (30 minutes per session, 5 sessions per week for 2 weeks).

Outcome measures included:

1. Visual Analog Scale (VAS): For pain intensity.
2. Oswestry Disability Index (ODI): For functional disability.
3. Pittsburgh Sleep Quality Index (PSQI): For sleep quality.
4. Epworth Sleepiness Scale (ESS): For daytime sleepiness. Assessments were performed at baseline (Day 0), Day 7, and Day 15 by trained physicians using standardized protocols. Data analysis employed mixed-effects linear regression models to evaluate treatment effects over time and between groups.

Ethical approval was obtained from the Ethics Committee of the Binh Dinh Hospital of Traditional Medicine and Rehabilitation and the Science and Technology Council of the Binh Dinh Department of Health (Approval Number: 445/QĐ-SYT).

This pilot study aims to provide preliminary clinical evidence on the efficacy and safety of intravascular photobiomodulation for pain and sleep management in chronic sciatica, serving as a foundation for larger-scale trials and contributing to the development of integrative, non-pharmacologic treatment strategies in rehabilitation medicine.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 18 years.
* Diagnosis of chronic sciatica pain lasting ≥ 3 months.
* Sleep disturbance defined by a Pittsburgh Sleep Quality Index (PSQI) score > 5.
* Pain intensity score ≥ 50 mm on a 100-mm Visual Analog Scale (VAS).
* Able to walk independently (with or without walking aids).
* Provided written informed consent to participate in the study.

Exclusion Criteria:

* Malignant diseases, autoimmune diseases, or systemic inflammatory disorders.
* History of prior spinal surgery.
* Acute low back pain of < 4 weeks' duration.
* Primary sleep disorders (e.g., narcolepsy, sleep apnea, circadian rhythm disorders).
* Diagnosed psychiatric conditions such as depression, anxiety, or delirium.
* Current use of psychotropic, antidepressant, hypnotic, corticosteroid, or antihistamine medications.
* Contraindications to low-level intravascular laser irradiation (e.g., hemophilia, acute myocardial infarction, acute stroke within 72 hours, active infection, pregnancy).
* Signs or suspicion of severe spinal conditions (e.g., cancer, vertebral fracture, spinal infection, or cauda equina syndrome).
* Concurrent involvement of lumbosacral nerve roots, plexus, or peripheral neuropathy confirmed by electrodiagnostic testing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index (PSQI) Score | Days 0 (baseline), 7, and 15 after initiation of treatment
  The Pittsburgh Sleep Quality Index (PSQI) is a self-reported questionnaire assessing sleep quality and disturbances over the previous month. It includes 19 items grouped into 7 components (subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction). Each component is scored from 0 to 3, and the global PSQI score ranges from 0 to 21, where higher scores indicate poorer sleep quality.

SECONDARY OUTCOMES:
Change in Visual Analog Scale (VAS) for Pain | Days 0, 7 and 15
  Pain intensity is measured using a 100-mm Visual Analog Scale (VAS), where 0 indicates "no pain" and 100 indicates "worst imaginable pain." Scores are categorized as follows: 0-1 (no pain), 1-4 (mild), 4-6 (moderate), >6 (severe). The change in VAS from baseline to each follow-up point will be analyzed.
Change in Oswestry Disability Index (ODI) | Days 0 (baseline), 7, and 15.
  The Oswestry Disability Index (ODI) is a standardized questionnaire that measures the degree of disability related to low back pain. It consists of 10 sections, each scored from 0 to 5. The total score is expressed as a percentage from 0% to 100%, where 0% indicates no disability and 100% indicates maximum disability. Higher scores represent worse functional impairment.
Change in Epworth Sleepiness Scale (ESS) Score | Days 0, 7, and 15
  The Epworth Sleepiness Scale (ESS) measures daytime sleepiness across eight daily situations, rated from 0 (no chance of dozing) to 3 (high chance of dozing). The total score ranges from 0 to 24, with higher scores indicating greater daytime sleepiness.

CONTACTS AND LOCATIONS:
Locations (1):
- Binh Dinh Traditional Medicine and Rehabilitation Hospital, Qui Nhon, Binh Dinh, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) that will be shared include: demographic characteristics (age, sex, BMI, occupation) and de-identified outcome data related to pain, sleep quality, disability, and daytime sleepiness (VAS, PSQI, ODI, ESS). No identifiable personal information will be shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: The de-identified individual participant data and supporting documents will be available upon publication of the main results and remain accessible for at least 3 years after study completion.
Access Criteria: Qualified researchers may request access to the data by submitting a written proposal and analysis plan to the principal investigator (Dr. Le Hoang Minh Quan, University of Medicine and Pharmacy at Ho Chi Minh City). Data will be shared after approval of the research proposal and execution of a data-sharing agreement ensuring compliance with confidentiality and ethical standards.

REFERENCES:
- See also: N. E. Adler and K. Newman (2002), "Socioeconomic disparities in health: pathways and policies", Health Aff (Millwood). 21(2), pp. 60-76. — https://pubmed.ncbi.nlm.nih.gov/11900187/
- See also: Daniel J Buysse, et al (1989), "The Pittsburgh Sleep Quality Index: a new instrument for psychiatric practice and research", J Psychiatry research. 28(2), pp. 193-213. — https://pubmed.ncbi.nlm.nih.gov/2748771/
- See also: J. C. Fu, N. K. Wang, Y. Y. Cheng and S. T. Chang (2022), "The Adjuvant Therapy of Intravenous Laser Irradiation of Blood (ILIB) on Pain and Sleep Disturbance of Musculoskeletal Disorders", J Pers Med. 12(8). — https://pubmed.ncbi.nlm.nih.gov/36013282/
- See also: Y. L. Chang and S. T. Chang (2022), "The effects of intravascular photobiomodulation on sleep disturbance caused by Guillain-Barré syndrome after Astrazeneca vaccine inoculation: Case report and literature review", Medicine (Baltimore). 101(6), e28758 — https://pubmed.ncbi.nlm.nih.gov/35147100/
- See also: S. Asih, et al. (2014), "Insomnia in a chronic musculoskeletal pain with disability population is independent of pain and depression", Spine J. 14(9), pp. 2000-7. — https://pubmed.ncbi.nlm.nih.gov/24333458/
- See also: Sirous Momenzadeh and et al (2015), "The intravenous laser blood irradiation in chronic pain and fibromyalgia", Journal of lasers in medical sciences. 6(1), pp. 6. — https://pmc.ncbi.nlm.nih.gov/articles/PMC4329142/